CLINICAL TRIAL: NCT06609733
Title: Comparative Effect of Clear Aligner Mandibular Advancement and Twin Block Appliances in Class II Malocclusion
Status: Completed | Type: Observational
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Lijun Tan, Associate Professor and Vice Director, Sichuan University
Other Study IDs: WCHS-IRB-CT-2023-195
Record Dates: First submitted 2024-09-16; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: CLASS II DIVISION 1 MALOCCLUSION
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- MA group: Patients receiving routine care for Class II malocclusion, which may include the use of Clear Aligner with Mandibular Advancement (MA) function appliances
  Interventions: Device: Clear aligner with mandibular function
- TB group: Patients receiving routine care for Class II malocclusion, which may include the use of Twin Block (TB) appliances
  Interventions: Device: Twin block

INTERVENTIONS:
Device: Twin block — The TB group used a single appliance continuously, with appropriate reduction of occlusal surface height by 1 mm when clinically indicated. Both groups had follow-up appointments every 6 weeks.
  Groups: TB group
Device: Clear aligner with mandibular function — The MA group underwent stepwise mandibular forward movement with clear aligners (Invisalign, Align Inc, CA, USA) worn for 22 hours/day and replaced every 7 days.
  Groups: MA group

SUMMARY:
The goal of this retrospective observational study is to compare the effects of Clear Aligner Mandibular Advancement (MA) and Twin Block (TB) appliances in treating Class II malocclusion, a condition where the lower jaw is underdeveloped. The main questions it aims to answer are:

1. Does mandibular advancement with clear aligners improve jaw and dental alignment as effectively as Twin Block appliances?
2. What are the differences in soft tissue changes, such as chin advancement and lip position, between these two treatments?

Researchers will compare MA and TB appliances to an untreated control group to evaluate their impact on skeletal, dental, and soft tissue outcomes. Participants in the study underwent cephalometric analysis (X-ray measurements) both before and after treatment to assess changes in jaw positioning, overbite, and overjet. The study focuses on how each treatment affects facial aesthetics and dental function.

Participants in the study will:

* Undergo treatment with either clear aligner mandibular advancement or Twin Block appliances.
* Attend follow-up appointments to monitor progress and assess treatment outcomes.

DETAILED DESCRIPTION:
Supplementary information for Study Design It was a retrospective study that collected patients' routine treatment X-rays (before and after treatment) to measure some angular and linear parameters from the X-rays.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed MA or TB treatment at the West China Hospital of Stomatology Orthodontic Department.
* Pretreatment lateral cephalometric radiographs showing cervical vertebral maturation stage (CVSM) II or III.
* Patients in the mixed dentition or early permanent dentition stages.
* Class II Division 1 malocclusion according to Angle's classification
* ANB angle > 4°; SNB ≤ 78°.
* Comprehensive medical records and necessary data available pre- and post-treatment.

Exclusion Criteria:

* Missing teeth, supernumerary teeth, or severe dental malformations affecting function.
* Poor oral hygiene.
* Systemic diseases or congenital deformities.
* History of dental or maxillofacial trauma.
* Incomplete or missing records.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of patients from the Orthodontics Department at West China Hospital of Stomatology, Sichuan University. This population includes individuals diagnosed with Class II malocclusion who are undergoing or have completed treatment with Mandibular Advancement (MA) or Twin Block (TB) appliances. Eligible participants for the treatment group are those in the mixed dentition or early permanent dentition stages, showing specific cephalometric characteristics such as an ANB angle greater than 4 degrees and an SNB angle less than or equal to 78 degrees.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Skeletal Measurements ( SNB angle) | Baseline and post-treatment cephalometric radiographs will be taken 1-2 weeks pre and 1-2 weeks post the 12-month treatment at West China School of Stomatology, Sichuan University.
  This study assesses skeletal changes in patients treated for Class II malocclusion with Twin Block (TB) or Mandibular Advancement (MA) appliances at West China School of Stomatology, Sichuan University. The evaluation focuses on the measurement of the SNB angle, a critical skeletal parameter, using cephalometric radiographs. These radiographs are taken as a routine part of the treatment to capture skeletal positioning before the treatment starts and after the treatment concludes. This allows for an analysis of the angular changes due to the orthodontic intervention, providing insights into the effectiveness of the appliances in correcting malocclusions.
Changes in Soft Tissue Measurements ( soft tissue chin thickness) | Baseline and post-treatment cephalometric radiographs will be taken 1-2 weeks pre and 1-2 weeks post the 12-month treatment at West China School of Stomatology, Sichuan University.
  This study assesses skeletal changes in patients treated for Class II malocclusion with Twin Block (TB) or Mandibular Advancement (MA) appliances at West China School of Stomatology, Sichuan University. The evaluation focuses on the measurement of the soft tissue chin thickness, using cephalometric radiographs. These radiographs are taken as a routine part of the treatment to capture skeletal positioning before the treatment starts (baseline) and after the treatment concludes (1-2 weeks post the 12-month treatment). This allows for an analysis of the angular changes due to the orthodontic intervention, providing insights into the effectiveness of the appliances in correcting malocclusions.
Changes in Skeletal Measurements (ANB angle) | Baseline and post-treatment cephalometric radiographs will be taken 1-2 weeks pre and 1-2 weeks post the 12-month treatment at West China School of Stomatology, Sichuan University.
  This study assesses skeletal changes in patients treated for Class II malocclusion with Twin Block (TB) or Mandibular Advancement (MA) appliances at West China School of Stomatology, Sichuan University. The evaluation focuses on the measurement of the ANB angle, a critical skeletal parameter, using cephalometric radiographs. These radiographs are taken as a routine part of the treatment to capture skeletal positioning before the treatment starts and after the treatment concludes. This allows for an analysis of the angular changes due to the orthodontic intervention, providing insights into the effectiveness of the appliances in correcting malocclusions.
Changes in Skeletal Measurements ( mandibular length) | Baseline and post-treatment cephalometric radiographs will be taken 1-2 weeks pre and 1-2 weeks post the 12-month treatment at West China School of Stomatology, Sichuan University
  This study assesses skeletal changes in patients treated for Class II malocclusion with Twin Block (TB) or Mandibular Advancement (MA) appliances at West China School of Stomatology, Sichuan University. The evaluation focuses on the measurement of the mandibular length (mm), a critical skeletal parameter, using cephalometric radiographs. These radiographs are taken as a routine part of the treatment to capture skeletal positioning before the treatment starts and after the treatment concludes. This allows for an analysis of the angular changes due to the orthodontic intervention, providing insights into the effectiveness of the appliances in correcting malocclusions.

CONTACTS AND LOCATIONS:
Locations (1):
- West China School of Stomatology, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
confidential

REFERENCES:
- [Background] Alsaggaf DH, Afify AR, Zawawi KH, Alsulaimani FF. Factors influencing the orthodontic treatment plan in Class II malocclusion. Am J Orthod Dentofacial Orthop. 2022 Jun;161(6):829-837.e1. doi: 10.1016/j.ajodo.2021.01.034. Epub 2022 Jan 29. PMID 35094890